CLINICAL TRIAL: NCT03102801
Title: A Study to Identify Biomarkers of Hypoglycaemia in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hull (Other)
Responsible Party: Principal Investigator, Thozhukat Sathyapalan, Professor, University of Hull
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Version 2
Record Dates: First submitted 2016-12-06; First posted 2017-04-06 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Type 2 Diabetes Mellitus With Hypoglycemia
MeSH Terms: interventions — Insulin, Regular, Human

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Type 2 diabetes arm (Active Comparator): Both arms will be subjected to Hypoglycaemia and compare results
  Interventions: Drug: Humulin S
- Non diabetics arm (Active Comparator): Both arms will be subjected to Hypoglycaemia and compare results
  Interventions: Drug: Humulin S

INTERVENTIONS:
Drug: Humulin S — Humulin S used to induce hypoglycaemia

SUMMARY:
Glucose is a sugar carried in the blood stream that body uses for energy. If someone has diabetes, blood glucose level can be erratic, sometimes becoming very low this is called Hypoglycaemia (or a "hypo"), and can happen when blood glucose levels drop below 4 mmol/l.

So far in order to prove that a hypo happened for a patient, blood glucose level can only be measured at time of the hypo and not after it.

In this study we are trying to identify certain chemical substances (biomarkers) in diabetic patients that may be measured in blood tests of the patient up to after 24 hours of the hypo and if we could prove that a hypo has happened we could adjust tablets and or insulin dosage in a way to prevent further hypos.

The study will be conducted in the Diabetes Centre in Hull Royal Infirmary and will involve three visits to the diabetes centre. The study can finish in a week time after the first visit.

Visit 1 is the screening visit to identify eligibility to take part in the study. Visit 2 insulin infusion will be given to make participants blood sugar level fall lower than normal for a short time and corrected quickly afterward. This is a stress for participant's body and should stimulate certain chemicals that we are trying to identify during hypo.

In Visit 3, the main purpose of this visit which is done 24 hours after insulin infusion is to take a blood sample and check how participants is after visit 2.

We will recruit 25 Type 2 Diabetic patients and 25 none diabetics to compare both results.

Both groups should not have ischemic heart disease, underactive thyroid or seizures and on stable dosage of medications.

DETAILED DESCRIPTION:
Background information It is well recognised that patients with both type 1 and type 2 diabetes suffering repeated hypoglycaemia are at risk of death and significant morbidity (1). This is of major clinical importance as currently, only the recording of a low blood sugar at the time of hypoglycaemia gives confirmation that a hypoglycaemic event has taken place. There are many instances when the confirmation or exclusion of a hypoglycaemic event would be beneficial.

Landmark studies such as the Diabetes Control and Complications Trial (DCCT) )(2) in type 1 diabetes and the in numerous large studies (UKPDS, ACCORD, ADVANCE, VADT(1, 3-7)) designed to look at whether intensive diabetes control in type 2 diabetes reduced microvascular and macrovascular cardiovascular events, have helped in establishing glycaemic targets which will contribute to preventing the development or worsening of retinopathy, nephropathy and neuropathy. What these studies exemplified was that as glycaemic control became stricter, the risk of hypoglycaemia increased (defined as a blood glucose fall to less than 3.9mmol/l according to American Diabetes Association guidelines)(1, 6, 7). For many patients, the main barrier to achieving optimal glycaemic targets to prevent complications are their increased risks of hypoglycaemia that remains the most feared complication of intensifying diabetes therapy for both patients and their health care professional.

Although hypoglycaemia has traditionally been considered a complication of the treatment for type 1 diabetes, it has recently been recognised as a problem in people with type 2 diabetes particularly those on intensive insulin therapy (8). In type 1 diabetes, patients on average experience two symptomatic events per week and one severe event, the latter of which is responsible for 2-4% of deaths. In type 2 diabetes the risk of a severe hypoglycaemic event is about 7% in the first few years following diagnosis rising to 25% thereafter. There are multiple concerns on the impact that a hypoglycaemic event may have leading to pathological, social and economic consequences. In the ACCORD study, the risk of death was significantly increased in those with one or more episode of severe hypoglycaemia in both the intensive and standard study treatment arms (1, 9). As plasma glucose falls to below 4.0mmol/L, a series of defensive response mechanisms occur, at individualised glycaemic thresholds, to reverse hypoglycaemia including a rise in catecholamine, cortisol and glucagon levels (10). This may lead to hypokalemia, prolonged QT interval, and cardiac arrhythmias (11). It may also lead to increased oxidative stress (12); impaired cardiovascular autonomic function for up to 16 hours afterwards (13); increased inflammatory markers (14); platelet activation (15) and promote vascular damage. These changes might be clinically relevant as hypoglycaemia was associated with cardiac ischemia (chest pain) when 72-h continuous glucose monitoring along with simultaneous cardiac Holter monitoring were performed in people with ischemic heart disease and type 2 diabetes treated with insulin (16). A few studies, in people with type 1 diabetes and healthy controls, suggested an increase in platelet activation with hypoglycaemia (15, 17) emphasising the increased risk that hypoglycaemia may have on cardiovascular events.

All of these changes may therefore result in the generation of biomarkers that may be able to identify the occurrence of a hypoglycaemia event after the blood glucose has reversed to normal or rebound hyperglycaemic levels have resulted. This will be of particular value in hypoglycaemic unawareness, nocturnal hypoglycaemia and events of uncertain aetiology where hypoglycaemia is part of the differential diagnosis.

An ability to determine whether a hypoglycaemic event has occurred through measurement of a biomarker will be of major impact for the confidence of patients and their healthcare providers allowing glycaemic control to be optimised and glycaemic targets to be reached through more stringent diabetes therapeutic treatment regimens.

The ability to identify nocturnal hypoglycaemia will be of particular value in all patients and will circumvent the need for continuous glucose monitoring or enforced waking at 3am to do blood glucose measurements that we currently have to rely on. Identification of biomarkers for hypoglycaemia will be of great value in the elderly population where it is often difficult to determine causes of, for example, feeling non specifically unwell, poor concentration, falls or faints, particularly as there are often multiple morbidities that are being treated at the same time (18).

From an economic perspective it is recognised that hypoglycaemia directly accounts for 95% of endocrine related emergency hospitalisations (19)and it is recognised that severe hypoglycaemia is associated with a total cost of around £2,152 (20) It can then be seen that a new method to determine hypoglycaemia through biomarker determination may help prevent severe hypoglycaemia by earlier recognition and prevent death and morbidity.

One promising biomarker is that of endothelial Microparticles which are heterogeneous population of vesicles playing a relevant role in the pathogenesis of vascular diseases, cancer and metabolic diseases such as diabetes mellitus.

They are released by virtually all cell types by shedding during cell growth, proliferation, activation, apoptosis or senescence processes.(21) Microparticles are consistently present in blood stream (22) they are the main regulators of cell to cell interactions, by carrying specific membrane antigens from their host cells, thereby acting as diffusible vectors in the trancellular exchange of biological information(23).

Microparticles expose membrane proteins of their mother cell for example CD31 is for endothelial cells and a proportion of platelets.(24) CD105,CD106, CD142, CD54, CD62E all Endothelial cells in nature.(25-28) An increased level of circulating Microparticles has been suggested to be one of the procoagulant determinants in patients with type 2 diabetes mellitus (29)Circulating levels of CD31+ (PECAM-1), CD105+, CD106+ and 62E+ endothelial-derived MPs as well as increased concentrations of fibrinogen+, tissue factor, P-selectin+ platelet-derived MPs have been shown to be significantly increased in T2DM patients as compared with non-diabetic controls (25, 26)Indeed, platelets of patients with T2DM are characterised by an hyperreactive phenotype with enhanced adhesion, aggregation, and activation(30), that may contribute to the pathogenesis of atherothrombotic complications(31-33). Therefore, high levels of specific endothelial and platelets Microparticles circulate in the blood of patients with atherosclerotic diseases, and can be used as biomarkers of vascular injury and potential predictors of cardiovascular outcome, especially in diabetic patients(34-37).

Aims and Objectives

Objectives :

Identification and comparison of Microparticles (CD105, CD106, CD31, CD54, CD62E, CD142) following a hypoglycemic event in patients with type 2 diabetes and in subjects without type 2 diabetes.

Study Design Prospective parallel study performed in the Diabetes research centre, Hull Royal Infirmary involving patients with type 2 diabetes and a control group without diabetes

ELIGIBILITY:
Inclusion Criteria for diabetic patients.

1. Men and women who are white British or white Europeans between 40 - 70 years of age with type 2 diabetes.
2. Duration of diabetes less than 10 years.
3. Stable dose of medication over the last 3 months.
4. No history of severe hypoglycemic in the preceding 3 months.
5. No hypoglycemic unawareness
6. Able to give informed consent.

Exclusion Criteria for diabetic patients.

1. Type 1 diabetes.
2. Duration of diabetes of more than 10 years.
3. Patients who are on insulin.
4. HbA1c of ≥ 10%.
5. BMI <18 or >50 kg/m2
6. Alcohol excess defined as 14 units per week for a man or a woman. Binge drinking is defined 6 units for a man or women in a single drinking session.
7. Renal impairment with estimated Glomerular Filtration Rate (eGFR<60 ml/min/1.73 m2).
8. Impaired Liver function tests defined as ALT or AST more than or equal 2.5 times upper limit of the normal.
9. History or presence of malignant neoplasms within the last 5 years( except basal and squamous cell skin cancer and in-situ carcinoma).
10. Psychiatric illness.
11. Any form of gastrointestinal tract surgery.
12. Any medications that can mask Hypoglycaemia such as B-Blockers or Clonidine.
13. Medication that may cause change in glucose metabolism.
14. Patients on any form of steroids in the last six months.
15. Female who is pregnant, breast feeding or intended to become pregnant or of child bearing potential not using adequate contraceptive methods.
16. History of pancreatitis (Acute or Chronic).
17. History of severe hypoglycaemia or hypoglycaemic unawareness.
18. Any disorder which in the opinion of the investigator might jeopardize subject's safety.
19. Contraindications to insulin infusion aiming for hypoglycaemia:

    * Ischaemic heart disease.
    * Epilepsy or previous history of seizures.
    * Drop attacks.
    * History of adrenal insufficiency.
    * Untreated hypothyroidism.

Inclusion Criteria for the control group.

1. Men and women who are white British or white Europeans between 40 - 70 years of age.
2. Stable dose of medications in last 3 months.
3. Able to give informed consent.

Exclusion Criteria for the control group

1. History of diabetes
2. BMI <18 or >50 kg/m2
3. HbA1C>6% (42mmol/mol)
4. Alcohol excess defined as 14 units per week for a man or a women. Binge drinking is defined 6 units for a man or women in a single drinking session.
5. Renal impairment with estimated Glomerular Filtration Rate (eGFR<60 ml/min/1.73 m2).
6. Impaired Liver function tests defined as ALT or AST more than or equal 2.5 times upper limit of the normal.
7. History or presence of malignant neoplasms within the last 5 years( except basal and squamous cell skin cancer and in-situ carcinoma).
8. Psychiatric illness
9. Female who is pregnant, breast feeding or intended to become pregnant or of child bearing potential not using adequate contraceptive methods.
10. Medication that may cause change in glucose metabolism
11. Any form of gastrointestinal tract surgery.
12. Patient on any form of steroids in the last 6 months.
13. Any disorder which in the opinion of the investigator might jeopardize subject's safety.
14. Contraindications to insulin infusion aiming for hypoglycaemia:

    * Ischaemic heart disease.
    * Epilepsy or previous history of seizures.
    * Drop attacks.
    * History of adrenal insufficiency.
    * Untreated hypothyroidism.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
Measurement of endothelial microparticles (composite number of CD105, CD106, CD142, CD54, CD62 & CD31) following hypoglycemic event | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hull and east Yorkshire Hospitals NHS Trust, Hull, United Kingdom

REFERENCES:
- [Derived] Moin ASM, Nandakumar M, Diboun I, Al-Qaissi A, Sathyapalan T, Atkin SL, Butler AE. Hypoglycemia-induced changes in complement pathways in type 2 diabetes. Atheroscler Plus. 2021 Nov 18;46:35-45. doi: 10.1016/j.athplu.2021.11.002. eCollection 2021 Dec. PMID 36643727
- [Derived] Ramanjaneya M, Bettahi I, Pawar K, Halabi NM, Moin ASM, Sathyapalan T, Abou-Samra AB, Atkin SL, Butler AE. MicroRNA Changes Up to 24 h following Induced Hypoglycemia in Type 2 Diabetes. Int J Mol Sci. 2022 Nov 24;23(23):14696. doi: 10.3390/ijms232314696. PMID 36499023
- [Derived] Moin ASM, Sathyapalan T, Atkin SL, Butler AE. The severity and duration of Hypoglycemia affect platelet-derived protein responses in Caucasians. Cardiovasc Diabetol. 2022 Oct 6;21(1):202. doi: 10.1186/s12933-022-01639-w. PMID 36203210
- [Derived] Ramanjaneya M, Priyanka R, Bensila M, Jerobin J, Pawar K, Sathyapalan T, Abou-Samra AB, Halabi NM, Moin ASM, Atkin SL, Butler AE. MiRNA and associated inflammatory changes from baseline to hypoglycemia in type 2 diabetes. Front Endocrinol (Lausanne). 2022 Aug 9;13:917041. doi: 10.3389/fendo.2022.917041. eCollection 2022. PMID 36017315
- [Derived] Nandakumar M, Moin ASM, Ramanjaneya M, Qaissi AA, Sathyapalan T, Atkin SL, Butler AE. Severe iatrogenic hypoglycaemia modulates the fibroblast growth factor protein response. Diabetes Obes Metab. 2022 Aug;24(8):1483-1497. doi: 10.1111/dom.14716. Epub 2022 May 3. PMID 35415885
- [Derived] Moin ASM, Nandakumar M, Al-Qaissi A, Sathyapalan T, Atkin SL, Butler AE. Potential Biomarkers to Predict Acute Ischemic Stroke in Type 2 Diabetes. Front Mol Biosci. 2021 Dec 1;8:744459. doi: 10.3389/fmolb.2021.744459. eCollection 2021. PMID 34926573
- [Derived] Butler AE, Al-Qaissi A, Sathyapalan T, Atkin SL. Angiopoietin-1: an early biomarker of diabetic nephropathy? J Transl Med. 2021 Oct 13;19(1):427. doi: 10.1186/s12967-021-03105-9. No abstract available. PMID 34645474
- [Derived] Atkin AS, Moin ASM, Nandakumar M, Al-Qaissi A, Sathyapalan T, Atkin SL, Butler AE. Impact of severe hypoglycemia on the heat shock and related protein response. Sci Rep. 2021 Aug 23;11(1):17057. doi: 10.1038/s41598-021-96642-8. PMID 34426634
- [Derived] Moin ASM, Al-Qaissi A, Sathyapalan T, Atkin SL, Butler AE. Soluble Neuropilin-1 Response to Hypoglycemia in Type 2 Diabetes: Increased Risk or Protection in SARS-CoV-2 Infection? Front Endocrinol (Lausanne). 2021 Jun 23;12:665134. doi: 10.3389/fendo.2021.665134. eCollection 2021. PMID 34248841
- [Derived] Moin ASM, Al-Qaissi A, Sathyapalan T, Atkin SL, Butler AE. Type 2 Diabetes Coagulopathy Proteins May Conflict With Biomarkers Reflective of COVID-19 Severity. Front Endocrinol (Lausanne). 2021 Jun 25;12:658304. doi: 10.3389/fendo.2021.658304. eCollection 2021. PMID 34248840
- [Derived] Moin ASM, Kahal H, Al-Qaissi A, Kumar N, Sathyapalan T, Atkin SL, Butler AE. Amyloid-related protein changes associated with dementia differ according to severity of hypoglycemia. BMJ Open Diabetes Res Care. 2021 Apr;9(1):e002211. doi: 10.1136/bmjdrc-2021-002211. PMID 33931404
- [Derived] Atkin AS, Moin ASM, Al-Qaissi A, Sathyapalan T, Atkin SL, Butler AE. Plasma heat shock protein response to euglycemia in type 2 diabetes. BMJ Open Diabetes Res Care. 2021 Apr;9(1):e002057. doi: 10.1136/bmjdrc-2020-002057. PMID 33879515
- [Derived] Moin ASM, Al-Qaissi A, Sathyapalan T, Atkin SL, Butler AE. Platelet Protein-Related Abnormalities in Response to Acute Hypoglycemia in Type 2 Diabetes. Front Endocrinol (Lausanne). 2021 Mar 30;12:651009. doi: 10.3389/fendo.2021.651009. eCollection 2021. PMID 33859620
- [Derived] Moin ASM, Sathyapalan T, Diboun I, Atkin SL, Butler AE. Identification of macrophage activation-related biomarkers in obese type 2 diabetes that may be indicative of enhanced respiratory risk in COVID-19. Sci Rep. 2021 Mar 19;11(1):6428. doi: 10.1038/s41598-021-85760-y. PMID 33742062
- [Derived] Moin ASM, Al-Qaissi A, Sathyapalan T, Atkin SL, Butler AE. Do biomarkers of COVID-19 severity simply reflect a stress response in type 2 diabetes: Biomarker response to hypoglycemia. Metabolism. 2021 Jan;114:154417. doi: 10.1016/j.metabol.2020.154417. Epub 2020 Nov 4. No abstract available. PMID 33157081
- [Derived] Moin ASM, Sathyapalan T, Atkin SL, Butler AE. Pro-fibrotic M2 macrophage markers may increase the risk for COVID19 in type 2 diabetes with obesity. Metabolism. 2020 Nov;112:154374. doi: 10.1016/j.metabol.2020.154374. Epub 2020 Sep 16. No abstract available. PMID 32949593